CLINICAL TRIAL: NCT01378494
Title: Bone Mineral Density in HIV+ Patients Recently Started on Antiretroviral Therapy (ART)
Brief Title: Bone Mineral Density in HIV+ Patients
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amy H. Warriner, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: F110105006
Record Dates: First submitted 2011-06-16; First posted 2011-06-22 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Osteoporosis
Keywords: osteoporosis; bone; HIV; antiretrovirals; inflammation
MeSH Terms: conditions — Osteoporosis; Inflammation

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV+: HIV+ patients that entered the 1917 Clinic at UAB as naive to ART

SUMMARY:
Utilizing an extremely well-characterized HIV cohort under observation as ART-naïve or since their first exposure to HIV treatment, the investigators will conduct a cross-sectional study with prospectively collected data to determine BMD in 200 subjects. Subjects identified were initially treatment naïve when entering the University of Alabama at Birmingham (UAB) 1917 HIV Clinic between 1999 and 2010; some have been under observation without being treated with ART therapy and others were newly started on ART therapy while under observation. For each subject, the investigators will determine associations between BMD and 1) cumulative viremia, 2) ART duration, and 3) ART type.

Hypothesis 1a: BMD will be lowest in HIV+ subjects with the highest levels of cumulative viremia.

Hypothesis 1b: BMD will be greatest in HIV+ persons with longest duration of ART therapy, after excluding those subjects treated with tenofovir.

Hypotheses 1c: BMD will be lower in subjects treated with tenofovir vs. other ART agents, after controlling for duration of therapy.

Additionally, the investigators will conduct a retrospective study in 100 patients HIV+ and were ART-naïve at the time of entry into the 1917 Clinic in whom the investigators will longitudinally evaluate the relationship between HIV viral load, inflammation, and bone turnover (through the measurement of HIV copy-years viremia, interleukin-6 {IL-6}, tumor necrosis factor alpha {TNF-a}, high-sensitivity c-reactive protein {hsCRP}, osteocalcin, and urine C-telopeptide {CTX}). The investigators will compare HIV patients at a similar stage of their disease who remain treatment naïve (either due to concerns for compliance or sufficient CD4 counts without treatment) (ART-) vs. those newly started on ART (ART+).

Hypothesis 2: Viral load, markers of inflammation, and markers of bone resorption will all decrease in ART+ vs. ART- persons.

DETAILED DESCRIPTION:
The life expectancy of persons infected with HIV has improved greatly since the institution of combination antiretroviral therapy (cART). However, many metabolic derangements have been discovered with long-term cART therapy, including lipodystrophy, insulin resistance, and, more recently, abnormal bone metabolism. It is well documented that bone mineral density (BMD) in HIV+ patients is lower when compared with the expected BMD in non-HIV patients [1-10]. The underlying cause of lower BMD is unknown but it is felt to be a multifactorial process [10-14]. Current guidelines recommend first line treatments consist of a combination of protease inhibitor (PI) or non-nucleoside reverse transcriptase inhibitor (NNRTI) in combination with two nucleoside reverse transcriptase inhibitors (NRTIs). Despite the known change in BMD in HIV+ persons, less is known about the effect of antiretroviral (ART) exposure and duration of treatment, ART type, and cumulative HIV viremia on bone health. This is demonstrated by studies showing loss of BMD with use of protease inhibitors compared to other regimen [15], other studies showing more detrimental effect from NRTIs [6, 9, 16], and yet others that have shown that BMD improves with all ART therapy [17]. Tenofovir (an NRTI), in particular, has been implicated as playing a role in bone changes, possibly due to its effect at the proximal tubule leading to a Fanconi-like syndrome with phosphate wasting [18]. Tenofovir led to significant reductions in BMD of children and this loss reversed after tenofovir was stopped [9]; other studies have shown similar deleterious effects [16]. A recent study evaluating the effect of continuous ART therapy vs. intermittent use for viral suppression showed that patients receiving continuous ART had greater loss of BMD, despite an increased risk of AIDS progression, myocardial infarction, or renal- or liver-failure [19]. However, prior longitudinal studies with longer follow-up have shown that the initial loss of BMD following ART is recovered and longer-term BMD changes are similar to changes seen in HIV-negative persons [20-22]. There is evidence that there is a positive correlation between HIV viremia and proinflammatory cytokines and that up-regulated proinflammatory cytokines may play a role in both osteoclast and osteoblast function. Prior studies have shown that during HIV infection osteoblast and osteoclast function is uncoupled and following ART treatment, regulation of bone turnover and formation ensues [23]. However, changes in cytokines have not been correlated with BMD and changes in bone turnover during routine ART treatment, to our knowledge. Most studies to date have been cross-sectional studies comparing HIV+ (with varying ART exposure histories) and HIV- persons or small longitudinal studies with limited sample sizes and short duration. It is not known if the decline of proinflammatory cytokines which occurs concurrent with the fall in HIV viral loads leads to improved regulation of bone formation and hence a lower rate of bone loss and lower risk of fracture.

ELIGIBILITY:
Inclusion Criteria:

* All treatment naïve patients seen in the 1917 Clinic between January 1, 1999 and December 31, 2010 will be identified.
* Of these patients, those who are currently under care at the time of the initiation of the study (>1 clinic visit in the past 12 months) will be eligible (regardless of current use of ART treatment).

Exclusion Criteria:

* Patients with a history of chronic renal failure (estimated GFR <30ml/min) will be excluded from the study.
* In addition, patients with a known diagnosis of a metabolic bone disease (i.e. osteoporosis, primary hyperparathyroidism, Paget Disease, Osteogenesis Imperfecta), multiple myeloma, cancer, untreated thyroid disease, or inflammatory bowel disease, or persons currently treated with or plans to begin an osteoporosis-specific medication (including estrogen) will be excluded from participation.
* Patients treated with oral glucocorticoids and anticonvulsants will also be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ART-naïve patients or patients followed since their first exposure to HIV treatment at the 1917 Clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | Baseline

SECONDARY OUTCOMES:
Pro-inflammatory and bone turnover markers | 6-12 months apart
  Change in IL-6, TNF-alpha, CRP, P1NP, Bone specific alkaline phosphatase, Serum NTX, and TRACP 5b at 6 and/or 12 months, as samples allow

CONTACTS AND LOCATIONS:
Overall Officials: Amy H Warriner, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States